CLINICAL TRIAL: NCT05680038
Title: A Real-world Study of Efficacy and Safety of Penpulimab in Maintenance Therapy in Patients With Post-transplant or Transplant-intolerant Lymphoma
Brief Title: Penpulimab in Maintenance Therapy in Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: WEI XU (Other)
Responsible Party: Sponsor-Investigator, WEI XU, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: Penp-001
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — penpulimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Penpulimab — Penpulimab is a modified PD1 inhibitor, which innovated the use of IgG1 subtype. On the basis of ensuring the stability of the antibody, it eliminated ADCC, ADCP, CDC and other effects that were not conducive to the efficacy of T cells and reduced the effect of ADCR by modifying the Fc segment

SUMMARY:
Panpulimab is a modified PD1 inhibitor, which innovated the use of IgG1 subtype. On the basis of ensuring the stability of the antibody, it eliminated ADCC, ADCP, CDC and other effects that were not conducive to the efficacy of T cells and reduced the effect of ADCR by modifying the Fc segment. There have been no studies on the safety and efficacy of Panpulimab in maintenance therapy after transplantation or in patients with transplant-intolerant lymphoma. The maintenance treatment of Panpulimab in our center has been preliminarily explored in clinic, and the results show good efficacy and safety. Therefore, based on the mechanism of PD1 monoclonal antibody maintenance therapy in lymphoma and the results of related clinical studies, this study proposed a regimen of peamprilizumab maintenance therapy for post-transplant or transplant intolerant lymphoma patients in real world studies, with the main purpose of observing the efficacy and safety of this regimen in lymphoma patients.

DETAILED DESCRIPTION:
After the completion of first-line induction and consolidation therapy, the lymphoma patients who received transplantation or were intolerant to transplantation were treated with Panpulimab monotherapy, 200 mg, once every three weeks, and were evaluated after six months of maintenance therapy. The patients who were evaluated as CR were excluded from the group, and the patients who did not reach CR were continued to take medication until CR. Review every 3 months from the first year of maintenance treatment and every 6 months from the second year to the fifth year.

ELIGIBILITY:
Inclusion Criteria:

1. Lymphoma patients who received transplantation or were intolerant to transplantation achieved remission after previous induction and consolidation therapy. Patients who were intolerant to transplantation here referred to lymphoma patients ≥60 years old or < 60 years old and recommended for transplantation by the guidelines;
2. Age ≥18 years old;
3. ECOG PS< 2 points;
4. Life expectancy is more than 3 months;
5. Patients were allowed to receive radiotherapy, but the last radiotherapy was given more than 7 days before the initial study drug administration;
6. Normal liver and kidney function, specific for direct bilirubin in serum, serum indirect bilirubin and/or cereal third transaminase, aspertate aminotransferase, serum creatinine 2 or less normal limit, creatinine clearance or ≥60 mL/min.
7. Normal bone marrow function, specific defined as absolute neutrophil count (ANC) acuity ≥1.0*10^9 / L, platelet ≥50 *10^9/L and ≥70 g/L or higher hemoglobin;
8. Women of childbearing age who used contraception or had a negative pregnancy test before enrollment, and who used contraception during the test period and within 8 weeks of the last drug administration; For men who were methodically contracepted or surgically sterilized during the trial period and 8 weeks after the last dose;
9. The subjects voluntarily joined the study and signed the informed consent with good compliance and follow-up.

Exclusion Criteria:

* 1. Pregnant or lactating women;

  2. Patients with a history of autoimmune diseases or syndromes requiring systemic use of steroid immunosuppressants, such as pituitaritis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.;

  3. The patient had received systemic glucocorticoids (prednisone > 20mg/ day) therapy (excluding nasal spray, inhaled or other topical corticosteroids) or any other form of immunosuppressive therapy;

  4. Uncontrolled heart disease, including unstable angina, acute myocardial infarction 6 months before randomization, congestive heart failure (NYHA) with a grade III or IV heart function; Or left ventricular ejection fraction < 50%;

  5. Known allergy to test drug ingredients;

  6. Patients receiving organ transplants;

  7. Has been diagnosed with or is undergoing treatment for a malignancy other than lymphoma, except for:
  * had received treatment for the purpose of cure, and had no malignancies with known active disease for ≥5 years prior to enrollment;

    * Well-treated basal cell carcinoma of the skin with no signs of disease (except melanoma);

      * Well-treated carcinoma in situ of the cervix with no signs of disease.

        8. Patients with grade 3 or above neurotoxic reactions in the two weeks prior to treatment;

        9. Severely infected persons;

        10. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study or the evaluation of the study results;

        11. Those who were considered unsuitable for inclusion by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma after transplantation or intolerant to transplantation
Sampling Method: Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the rates of PFS in 2-years | 24 months
  the rates of PFS in 2-years

SECONDARY OUTCOMES:
the rates of OS in 2-years | 24 months
  the rates of OS in 2-years
CR | 24 months
  CR
the rate of CR converted from PR | 24 months
  the rate of CR converted from PR
Number of participants with treatment-related Adverse Events and Serious Adverse Events as assessed by NCI-CTC 5.0 | 24 months
  AE and serious adverse events (SAEs) were observed and graded according to NCI-CTC version 5.0

IPD SHARING:
Plan to Share IPD: Undecided